CLINICAL TRIAL: NCT07089615
Title: Prospective, Open Label, Pivotal Study of the Accuracy of the CapsoCam® Colon (CV-3) in Detecting Colonic Polyps, Using Colonoscopy as the Reference
Brief Title: Prospective, Open-label, Non-significant Risk, Multicenter Study Comparing the Polyp Detection of the Study Device to That of the Colonoscopy Reference
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLN-CVI-5794 2nd Generation
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- A new capsule design is being used from that of the first phase of the study. (Experimental)
  Interventions: Device: Capsule swallow

INTERVENTIONS:
Device: Capsule swallow — Participant will swallow the investigational device

SUMMARY:
Note: This is the same study protocol as NCT04607746 with slight changes to how the videos will be read and a 2nd generation capsule is being studied.

The purpose of this study is to evaluate the safety and effectiveness of CapsoCam® Colon (CV-3) endoscope system for the detection of colonic polyps and to show that AI-based CADe improves the polyp-detection accuracy and efficiency of capsule video readers. It will use colonoscopy results as a reference.

The participant will:

1. prep for and swallow a study capsule and then
2. prep for and undergo a colonoscopy either the following day or 3-6 weeks later

ELIGIBILITY:
Inclusion Criteria:

1. 45-75 years of age
2. Committed to undergo a colonoscopy.
3. Choose to participate and must have signed the IRB-approved informed consent document and agreed to release colonoscopy images and results report to Sponsor

Exclusion Criteria:

1. Colonoscopy or CT-colonography within the past 5 years that demonstrated no polyps
2. Has contraindication for capsule endoscopy or colonoscopy
3. Subject is suspected or diagnosed with familial adenomatous polyposis, hereditary non polyposis colon cancer, or any high-risk genetic syndrome
4. Subject is suspected or diagnosed with inflammatory bowel disease such as ulcerative colitis or Crohn's disease
5. History of incomplete colonoscopy
6. Type I or uncontrolled II Diabetes (Uncontrolled defined as HbA1C>6.4 within the past 3 months and/or with history of constipation or gastroparesis).
7. Impaired cardiac function assessed as greater than NYHA Class II
8. History of small- or large-bowel obstructive condition
9. Known history of swallowing disorder, and/or ischemic bowel disease neuropathies and/or radiation enteritis
10. Known history of NSAID enteropathy and stricture resulting from taking NSAIDs on a regular basis that, in the opinion of the Investigator, would put the subject at greater risk for capsule endoscope retention
11. Known allergy to ingredients used in bowel preparation and boosters
12. Daily and/or regular narcotic use
13. Decompensated cirrhosis
14. Prior abdominal radiation therapy
15. Diagnosis of anorexia or bulimia
16. History of or suspicion of any of the following: strictures, volvulus or intestinal obstruction, or internal hernias or abdominal surgeries that the Investigator believes should exclude the patient from study participation
17. Known or suspected megacolon
18. Scheduled to undergo MRI examination within 7 days after ingestion of the capsule
19. Has known slow gastric-emptying time or confirmed diagnosis of gastroparesis
20. Pregnant or nursing or of child-bearing potential and does not agree to practice medically acceptable methods of contraception. Women of child bearing potential (WOCBP) must have a negative urine pregnancy test at screening.
21. Unable to follow or tolerate fasting, bowel preparation, and other study procedures
22. Any documented medical or psychological condition or significant concurrent illness which, in the Investigator's opinion, would make it unsafe for the subject to participate in this research study or would affect the validity of the study results
23. Are currently enrolled in an interventional clinical study or currently enrolled in or within the last 30 days, a pharmaceutical clinical study
24. Chronic constipation as defined by <3 bowel movements per week, or the use of routine laxatives (other than fiber) to attain regular bowel movements

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Positive Percentage Agreement | From capsule swallow to Colonoscopy - up to 6 weeks
  • Positive Percent Agreement (PPA) of the study device with computer assisted detection (CADe) for detecting the presence in a subject of the largest polyp detected by optical colonoscopy (OC) if that polyp is ≥ 6 mm, where a match is considered to have occurred if a polyp detected by the device is assessed as having a size within plus or minus 50% of the size of the polyp detected by OC and as having a location within the same or an adjacent colon segment.
Negative Percentage Agreement | From Capsule swallow to colonoscopy - Up to 6 weeks
  • Negative percent agreement (NPA) of the study device with CADe for not detecting any polyp ≥ 6 mm in a subject for whom OC did not detect any polyp ≥ 6 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Suejin Kim Study PI, M.D., Principal Investigator
Locations (11):
- United States (11):
  - SB Gastro Clinical Research, Chula Vista, California
  - Gastro Care Institute, Lancaster, California
  - Knowledge Research Center, Orange, California
  - Advanced Research Institute, St. Petersburg, Florida
  - Digestive Health Services, Downers Grove, Illinois
  - Gastroenterology and Internal Medicine Specialists, Lake Barrington, Illinois
  - Northshore Center for Gastroenterology, Libertyville, Illinois
  - Suburban Gastroenterology, Naperville, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Gastroenterology Group of Rochester, Rochester, New York
  - Great Lakes Gastroenterology Research, Mentor, Ohio

IPD SHARING:
Plan to Share IPD: No